CLINICAL TRIAL: NCT06402006
Title: A Comparative Study Between Ultrasound Guided Erector Spinae Plane Block and Combined Ultrasound Guided Pericapsular Nerve Group (PENG) and Lateral Femoral Nerve Block Following Total Hip Arthroplasty
Brief Title: A Comparative Study Between Ultrasound Guided Erector Spinae Plane Block and Combined Ultrasound Guided Pericapsular Nerve Group and Lateral Femoral Nerve Block Following Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, riham fathy galal, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FAMSU R79/2024
Record Dates: First submitted 2024-04-28; First posted 2024-05-07 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined hip joint PENG block and LFCN block (Experimental): Combined hip joint pericapsular nerve group block(PENG) and lateral femoral cutaneous nerve block
  Interventions: Procedure: PENG block; Procedure: LFCN block
- ESP block (Experimental): Erector spinae plane block(ESP)
  Interventions: Procedure: ESP block

INTERVENTIONS:
Procedure: PENG block — pericapsular nerve group block
  Arms: Combined hip joint PENG block and LFCN block
Procedure: LFCN block — Lateral femoral cutaneous nerve block
  Arms: Combined hip joint PENG block and LFCN block
Procedure: ESP block — Erector spinae plane block
  Arms: ESP block

SUMMARY:
The patients will be randomized into 2 equal groups by a computer-generated random numbers table, named group A, B.

Group A: patients will receive Pericapsular nerve group block and lateral femoral cutaneous nerve blocks.

Group B: Patients will receive Erector spinae plane block.

After IV access insertion and oxygen nasal cannula application, monitoring will be applied for all patients, sedation in the form of midazolam 0.02mg/kg with or without fentanyl 0.5-1 mcg/kg will be administered to any of the patients who felt discomfort or could not tolerate the procedure.

For (Group A) PENG block will be done before spinal anesthesia.

LFCN block will be performed.

For (Group B), ESP block will be done before spinal anesthesia.

Spinal anesthesia will be chosen as the main anesthetic technique.

In postoperative period all patients will receive the same adjuvant multimodal analgesia which will be 1000 mg of paracetamol with or without 30 mg ketorolac depending on comorbidities and depending on the patients" needs.

DETAILED DESCRIPTION:
The patients will be randomized into 2 equal groups by a computer-generated random numbers table, named group A, B.

Group A: patients will receive PENG and LFCN blocks.

Group B: Patients will receive ESP block, which will be the control group.

After obtaining approval from Ain Shams hospital academic and ethical committee, written, informed and valid consent will be taken from all participants after proper explanation of the study procedure and the expected outcome in a clear language for patients of either sex, aging from 18 to 65 years old, ASA physical status (I, II) scheduled for total hip arthroplasty surgeries.

Patients with the following criteria will be excluded from the study: Patient refusal, ASA physical status III or more, known allergy to any of the study drugs, infection at the site of injection, history of cardiovascular, renal, hepatic or neuromuscular diseases, history of any psychiatric disorder, presence of any coagulopathy, chronic opioid, gabapentin or pregabalin use, BMI more than 35 kg/m2. Patients will be randomly assigned to either both PENG and LFCN blocks and ESP block with ultrasound guidance before spinal anesthesia.

After IV access insertion and oxygen nasal cannula application, ECG (Electrocardiography), pulse oximeter, noninvasive blood pressure monitoring will be applied for all patients, sedation in the form of midazolam 0.02mg/kg with or without fentanyl 0.5-1 mcg/kg will be administered to any of the patients who felt discomfort or could not tolerate the procedure.

For (Group A) PENG block will be done before spinal anesthesia ultrasound-guided using a curvilinear array ultrasound transducer (2-5 MHz) Sono site M-turbo ultrasonography. While the patient is in the supine position, the probe will be placed in parallel to the inguinal crease and will be rotated clockwise until visualizing femoral artery, iliopsoas muscle tendon, anterior inferior iliac spine (AIIS) and ilio-pubic eminence. 22G 80 mm needle will be inserted in plane from lateral side of probe until tip of needle touch iliopubic eminence, after negative aspiration 20 ml of bupivacaine 0.5% will be injected. Success of injection will be confirmed by fluid spreading between the iliopsoas tendon and periosteum of iliopubic eminence.

LFCN block will be performed using linear ultrasound probe (10-15 MHz). while the patient is in supine position the probe will be directed caudally to AIIS until visualizing LFCN between sartorius muscle and tensor fascia latae. 5 ml of bupivacaine will be injected after negative aspiration.

For (Group B), ESP block will be done before spinal anesthesia in the lateral decubitus position by curvilinear probe (2-5 MHz). Probe will be placed on the third lumber vertebra in the parasagittal line to identify the transverse process of L3. Needle will be directed in plane caudo-cephalic to the lateral edge of L3 transverse process. 30 ml of bupivacaine will be injected under visualization along the erector spinae plane. Correct placement will be defined by spread of local anesthetic cranially and caudally from injection point, dissecting the plane between the transverse processes and erector spinae muscles.

Spinal anesthesia will be chosen as the main anesthetic technique by injecting 3-3.5 ml of hyperbaric bupivacaine 0.5% by 24 G pencil-point needle at L2-L3 or L3-L4 space with 25 ug of fentanyl as adjuvant while patient is in setting position.

In postoperative period all patients will receive the same adjuvant multimodal analgesia which will be 1000 mg of paracetamol with or without 30 mg ketorolac depending on comorbidities and depending on the patients" needs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of anesthesiologists' physical status (ASA) I to III.
2. Aged 18 to 65 years.
3. Both sexes.
4. Patients scheduled for total hip arthroplasty.

Exclusion Criteria:

1. Patient refusal
2. ASA physical status III or more.
3. Patients with known allergy to any of the study drugs.
4. Infection at the site of injection.
5. Patients with history of cardiovascular disease.
6. Patients with renal disease.
7. Patients with hepatic disease.
8. Patients with neuromuscular disease.
9. Presence of any coagulopathy.
10. Chronic opioid, gabapentin or pregabalin use.
11. Patients with history of any psychiatric disorder.
12. BMI more than 35 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
individual visual analog pain scores at 0, 6, 12, 24 and 48 h postoperatively (VAS; 0 = no pain and 10 = worst pain imaginable). | 48 hours
  The primary outcomes include : individual visual analog pain scores at 0, 6, 12, 24 and 48 h postoperatively (VAS; 0 = no pain and 10 = worst pain imaginable).
presence of moderate-to-severe pain, defined as pain score 4 or greater during the first 48 h postoperative. | 48 hours
  presence of moderate-to-severe pain, defined as pain score 4 or greater during the first 48 h postoperative.
analgesic consumption in post-anesthesia care unit, and during the first 48 h post-surgery (converted to IV pethidine equivalents). | 48 hours
  analgesic consumption in post-anesthesia care unit, and during the first 48 h post-surgery (converted to IV pethidine equivalents).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university hospitals, Cairo, Egypt